CLINICAL TRIAL: NCT01322490
Title: A Randomized, Double-blind, Phase 3 Efficacy Trial of PROSTVAC-V/F +/- GM-CSF in Men With Asymptomatic or Minimally Symptomatic Metastatic Castrate-Resistant Prostate Cancer
Acronym: Prospect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNIT-PRV-301
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer Metastatic
Keywords: PROSTVAC; metastatic; prostate cancer; castrate-resistant; vaccine; immunotherapy; Phase 3
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — PROSTVAC; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PROSTVAC-V/F-TRICOM + GM-CSF (Experimental): * PROSTVAC-V-TRICOM
  * PROSTVAC-F-TRICOM
  * GM-CSF
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Drug: GM-CSF
- PROSTVAC-V/F-TRICOM + GM-CSF placebo (Experimental): * PROSTVAC-V-TRICOM
  * PROSTVAC-F-TRICOM
  * GM-CSF placebo
  Interventions: Biological: PROSTVAC-V; Biological: PROSTVAC-F; Other: GM-CSF Placebo
- Placebo Control (Placebo Comparator): PROSTVAC V/F Placebo + GM-CSF Placebo
  Interventions: Other: GM-CSF Placebo; Biological: Placebo

INTERVENTIONS:
Biological: PROSTVAC-V
  Arms: PROSTVAC-V/F-TRICOM + GM-CSF; PROSTVAC-V/F-TRICOM + GM-CSF placebo
Biological: PROSTVAC-F
  Arms: PROSTVAC-V/F-TRICOM + GM-CSF; PROSTVAC-V/F-TRICOM + GM-CSF placebo
Drug: GM-CSF
  Arms: PROSTVAC-V/F-TRICOM + GM-CSF
Other: GM-CSF Placebo
  Arms: PROSTVAC-V/F-TRICOM + GM-CSF placebo; Placebo Control
Biological: Placebo — PROSTVAC V/F Placebo
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine whether PROSTVAC alone or in combination with GM-CSF is effective in prolonging overall survival in men with few or no symptoms from metastatic, castrate-resistant prostate cancer.

DETAILED DESCRIPTION:
BNIT-PRV-301 is a randomized, placebo-controlled, multi-center, global Phase 3 efficacy trial of PROSTVAC in men with asymptomatic or minimally symptomatic, metastatic, castrate-resistant prostate cancer. It is a 3-arm study and will evaluate overall survival in two separate comparisons, PROSTVAC plus adjuvant dose GM-CSF versus controls, and PROSTVAC without GM-CSF versus controls.

Patients will be randomized with equal probability into one of three double-blind arms. The intended interventions for randomized patients are:

1. (Arm V+G) PROSTVAC-V/F plus adjuvant dose GM-CSF
2. (Arm V) PROSTVAC-V/F plus GM-CSF placebo
3. (Arm P) Double placebo

ELIGIBILITY:
Inclusion Criteria:

Men, ≥18years of age with documented asymptomatic or minimally symptomatic metastatic castration-resistant prostate cancer.

Documented progressive disease post surgical castration or during androgen suppression therapy, or during complete androgen blockade therapy and withdrawal. Documented by either criterion a (Radiological progression), OR criterion b (PSA progression).

1. Radiological progression defined as any new/enlarging bone metastases or new/enlarging lymph node disease, consistent with prostate cancer.

   OR
2. PSA progression defined by sequence of rising values separated by > 1 week (2 separate increasing values) over a threshold minimum of 2.0 ng/ml. (PCWG2 PSA eligibility criteria).

Chemotherapy naïve and Vaccinia-experienced (previous smallpox vaccination). Currently using a GnRH agonist or antagonist (unless surgically castrated).

Exclusion Criteria:

Cancer-related pain requiring scheduled opioid narcotics for control (as needed, ≤ 2x per week is allowed).

Metastasis to organ systems other than lymph nodes and/or bone. Estimated PSA doubling time of <1 month as established within 6 months of the anticipated first dose of vaccine or placebo.

Concurrent or prior Provenge (sipuleucel-T) immunotherapy for prostate cancer. Receipt of an investigational agent within 30 days (or 60 days for an antibody-based therapy) of the first planned dose of PROSTVAC-V/F.

History of prior malignancies other than prostate cancer within the past 3 years, excluding successfully resected basal or squamous cell carcinoma of the skin.

Congestive heart failure (NYHA Class II, III, or IV), unstable angina, ventricular or hemodynamically significant atrial arrhythmia, or cardiovascular disease such as stroke or myocardial infarction (current or within the past 6 months) Confirmed positive for HIV, hepatitis B, and /or hepatitis C. Immunodeficiency or splenectomy. History of or active autoimmune disease, persons with vitiligo are not excluded. Diabetics are not excluded if the condition is well controlled.

History of atopic dermatitis or active skin condition (acute, chronic, exfoliative) that disrupts the epidermis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1297 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L. Gulley, MD, Principal Investigator — National Cancer Institute (NCI); Philip Kantoff, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (220):
- United States (84):
  - Alaska Clinical Research Center, Llc, Anchorage, Alaska
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - Desert Hematology-Oncology, Rancho Mirage, California
  - San Bernardino Urological Associates, San Bernardino, California
  - San Diego Clinical Trials, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Stanford Advanced Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Manatee Medical Research Institute, LLC, Bradenton, Florida
  - Florida Urology Physicians, Fort Myers, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - James A Haley Veteran Affairs Medical Center, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Jesse Brown VA, Chicago, Illinois
  - First Urology PSC, Jeffersonville, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - The Iowa Clinic, PC Iowa Urology, West Des Moines, Iowa
  - Tulane University, New Orleans, Louisiana
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Maryland Prostate Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - National Cancer Institute - Center for Cancer Research, Bethesda, Maryland
  - Myron Murdock M.D. LLC, Greenbelt, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City VA Medical Center, Kansas City, Missouri
  - GU Research Network, LLC, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - VA Sierra Nevada HealthCare System, Reno, Nevada
  - Delaware Valley Urology LLC - Westhampton, Mount Laurel, New Jersey
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Brooklyn Urology Research Group, Brooklyn, New York
  - University Urology Associates, New York, New York
  - Hudson Valley Urology, P.C., Poughkeepsie, New York
  - Presbyterian Hospital Center for Cancer Research, Charlotte, North Carolina
  - Northeast Urology Research, Concord, North Carolina
  - Regional Cancer Care PA, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - W.G. (Bill) Hefner VA Medical Center, Salisbury, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Urology Research, Columbus, Ohio
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Urologic Consultants of Southeaster PA LLP, Bala-Cynwyd, Pennsylvania
  - Urological Associates Of Lancaster, Lancaster, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Ralph H Johnson VAMC, Charleston, South Carolina
  - WJB Dorn VA Medical Center, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of TN Medical Center, Knoxville, Tennessee
  - The West Clinic, P.C., Memphis, Tennessee
  - James H. Quillen Veterans Affairs Medical Center, Mountain Home, Tennessee
  - Urology Associates, PC, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Central Texas Veterans Health Care System, Temple, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - White River Junction Veterans Affairs Medical Center, White River Junction, Vermont
  - Virginia Oncology Associates PC, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - The Schiffler Cancer Center, Wheeling, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (10):
  - Sydney Haematology and Oncology Clinic, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Monash Medical Centre - Moorabbin Campus, Bentleigh East
  - Barwon Health, Geelong
  - St John of God Hospital, Subiaco
  - Border Medical Oncology, Wodonga
  - Princess Alexandra Hospital, Woolloongabba
- Belgium (6):
  - Ziekenhuisnetwerk Antwerpen - AZ Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
  - H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Canada (11):
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Capital District Health Authority, Halifax, Nova Scotia
  - Brantford Urology Research, Brantford, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - St. Josephs Healthcare Hamilton Research Ethics Board, Hamilton, Ontario
  - Queen's University at Kingston, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Female/Male Health Centres, Oakville, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec Hotel Dieu, Québec
- Denmark (7):
  - Aalborg Sygehus, Aalborg
  - Skejby Sygehus, Århus N
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Herlev Hospital, Herlev
  - Holstebro Sygehus, Holstebro
  - Storstrømmens Sygehus Næstved, Næstved
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (13):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Départemental La Roche sur Yon, Luçon, Montaigu - Les Oudaries, La Roche-sur-Yon
  - Centre Léon Bérard - Centre régional de lutte contre le cancer Rhône-Alpes, Lyon
  - Centre d'Oncologie de Gentilly, Nancy
  - HIA du Val de Grâce, Paris
  - Institut Curie, Paris
  - Fondation Hôpital Saint-Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot - Centre de lutte contre le cancer, Reims
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Hôpital Bretonneau, Tours
  - Centre Alexis Vautrin - Centre Régional de lutte contre le cancer de Lorraine, Vandœuvre-lès-Nancy
- Germany (14):
  - Stadtisches Klinikum Muchen GmbH, Munich, Bavaria
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann-Wolfgang-Goethe-Universität Frankfurt am Main, Frankfurt
  - Chirurgische Universitätsklinik Freiburg, Freiburg im Breisgau
  - Martini-Klinik am UKE GmbH, Hamburg
  - Klinikum der Friedrich-Schiller-Universität Jena, Jena
  - Universitätsmedizin der JGU Mainz, Mainz
  - Klinikum der Philipps-Universität Marburg, Marburg
  - Studienpraxis Urologie, Reutlingen
  - Universitätsklinikum Tübingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Landspitali University Hospital, Reykjavik, Iceland
- Israel (7):
  - Soroka University Medical Center, Beersheba
  - Bnei Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Assaf Harofe Medical Center, Tzrifin
- Netherlands (5):
  - NKI-AVL, Amsterdam
  - VUMC, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
- Poland (5):
  - AMEDS CENTRUM Sp. z o.o., Grodzisk Mazowiecki
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Szpital sw Elzbiety - Mokotowskie Centrum Medyczne Sp. z o. o., Warsaw
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - Klinika Urologii i Onkologii Urologicznej, Uniwersytecki Szpital Kliniczny we Wrocławiu, Wroclaw
- Puerto Rico (2):
  - Ponce School of Medicine, Ponce
  - Alliance for Research and Knowledge, San Juan
- Russia (15):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Kazan State Medical University, Kazan'
  - Moscow Research Oncology Institute n.a. P.A.Gertsen, Moscow
  - Clinical Oncology Dispensary, Omsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Orel Oncology Center, Oryol
  - St. Petersburg Medical Academy of Postgraduate Education, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - "Clinic Andros" LLC, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - "Orkli" LLC, Saint Petersburg
  - Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - Regional Clinical Oncology Center, Vladimir
  - Regional Clinical Oncology Hospital, Yaroslavl
- Spain (23):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital 12 de Octubre, Madrid, Madrid, Communidad de
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Hospital Vall D´Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital General Universitario Gregorio Marañon, Madrid
  - MD Anderson International Espana, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Althaia: Xarxa Assistencial de Manresa, Manresa
  - Hospital General Carlos Haya, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Fundación Hospital Manacor, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Virgen del Rocio, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (14):
  - Bristol Haematology & Oncology Centre, Bristol, UK
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Velindre Hospital, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University of Surrey, Guildford
  - Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds
  - St Bartholomews Hospital, London
  - The Royal Marsden, London
  - St Mary's Hospital, London
  - Christie Hospital, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Plymouth Hospitals NHS Trust, Derriford Hospital, Plymouth
  - University of Southampton, Southampton
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Gulley JL, Borre M, Vogelzang NJ, Ng S, Agarwal N, Parker CC, Pook DW, Rathenborg P, Flaig TW, Carles J, Saad F, Shore ND, Chen L, Heery CR, Gerritsen WR, Priou F, Langkilde NC, Novikov A, Kantoff PW. Phase III Trial of PROSTVAC in Asymptomatic or Minimally Symptomatic Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2019 May 1;37(13):1051-1061. doi: 10.1200/JCO.18.02031. Epub 2019 Feb 28. PMID 30817251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 3, randomized, placebo-controlled, multicenter, multi-country efficacy trial of PROSTVAC administered SC to adult males with asymptomatic mCRPC, and was designed to enroll approximately 1200 men. Subjects were randomly assigned with equal probability (1:1:1) to one of three double-blind treatment arms.
Pre-assignment Details: Screening activities were completed within 28 days prior to the first dose of any medication and were completed prior to dosing. Subjects who required anti-androgen wash-out specifically for this protocol were consented prior to beginning withdrawal of therapy, however, no other screening procedures were performed the subject was deemed eligible.
Groups:
- PROSTVAC-V/F-TRICOM + GM-CSF Placebo: PROSTVAC V/F + Placebo GM-CSF, where PROSTVAC V is given SC at 2x10^8 Inf.U/0.5mL (Day 1) and PROSTVAC F is given SC at 1x10^9 Inf.U/0.5mL (Weeks 3, 5, 9, 13, 17, 21). Placebo GM-CSF was saline for injection (on days of PROSTVAC injection and three subsequent days).
- PROSTVAC-V/F-TRICOM + GM-CSF: PROSTVAC V/F + GM-CSF, where PROSTVAC V is given SC at 2x10^8 Inf.U/0.5mL (Day 1) and PROSTVAC F is given SC at 1x10^9 Inf.U/0.5mL (Weeks 3, 5, 9, 13, 17, 21). GM-CSF is given SC at 100ug (on days of PROSTVAC injection and three subsequent days).
- Placebo Control: Placebo PROSTVAC V/F + Placebo GM-CSF, where Placebo PROSTVAC V/F is an empty fowlpox vector (Day 1, Weeks 3, 5, 9, 13, 17, 21). Placebo GM-CSF was saline for injection (on days of PROSTVAC injection and three subsequent days).
Period: Treatment Period
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control
Started | 432 | 432 | 433
Treated | 429 | 429 | 428
Completed | 300 | 279 | 280
Not Completed | 132 | 153 | 153
Not completed — Adverse Event | 12 | 18 | 15
Not completed — Death | 5 | 7 | 3
Not completed — Lack of Efficacy | 89 | 100 | 112
Not completed — Physician Decision | 0 | 2 | 1
Not completed — Protocol Violation | 7 | 5 | 4
Not completed — Withdrawal by Subject | 14 | 16 | 11
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Other per report | 2 | 2 | 1
Not completed — Randomized but Not Treated | 3 | 3 | 5
Period: Long Term Follow-up Period
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control
Started | 409 (You did not have to complete treatment to enter follow up.) | 408 (You did not have to complete treatment to enter follow up.) | 413 (You did not have to complete treatment to enter follow up.)
Completed | 0 | 0 | 0
Not Completed | 409 | 408 | 413
Not completed — Death | 235 | 239 | 236
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Withdrawal by Subject | 9 | 6 | 6
Not completed — Study Terminated by Sponsor | 160 | 158 | 165
Not completed — Other per report | 3 | 2 | 2
Not completed — Unknown/Missing | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat, including all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control | Total
Number analyzed (Participants) | 432 | 432 | 433 | 1297
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 104 | 121 | 109 | 334
  >=65 years | 328 | 311 | 324 | 963
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.00) | 70.6 (8.42) | 71.4 (8.33) | 71.1 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 432 | 432 | 433 | 1297
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 18 | 40
  Not Hispanic or Latino | 418 | 421 | 415 | 1254
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 7 | 6 | 7 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 17 | 25 | 23 | 65
  White | 404 | 400 | 403 | 1207
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 2 | 1 | 2 | 5
  United States | 124 | 141 | 129 | 394
  United Kingdom | 31 | 29 | 39 | 99
  Iceland | 4 | 3 | 3 | 10
  Russia | 50 | 52 | 61 | 163
  Spain | 45 | 33 | 48 | 126
  Canada | 30 | 13 | 26 | 69
  Netherlands | 6 | 4 | 6 | 16
  Belgium | 12 | 8 | 10 | 30
  Denmark | 34 | 42 | 32 | 108
  Poland | 6 | 9 | 5 | 20
  Israel | 13 | 11 | 5 | 29
  Australia | 36 | 38 | 27 | 101
  France | 29 | 28 | 28 | 85
  Germany | 3 | 13 | 6 | 22
  Estonia | 7 | 7 | 6 | 20
Randomization Stratum [Count of Participants; unit: Participants] — Randomization stratum based on PSA 50ng/mL cut and LDH 200 U/L cut at baseline.
  Participants
    PSA < 50 ng/mL and LDH < 200 U/L | 168 | 168 | 168 | 504
    PSA < 50 ng/mL and LDH >= 200 U/L | 135 | 135 | 135 | 405
    PSA >= 50 ng/mL and LDH < 200 U/L | 65 | 64 | 64 | 193
    PSA >= 50 ng/mL and LDH >= 200 U/L | 64 | 65 | 66 | 195

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The time between the date of randomization and the date of death due to any cause. Subjects who did not experience death or the competing events of "definite" loss to follow-up or withdrawal of consent were right censored at the date of last contact. OS was calculated using the formula: OS = Date of death/competing event/censoring - date of randomization + 1.
Time Frame: Randomization through the date of death due to any cause. Subjects were followed up for approximately 6 years from the first subject randomized to the completion of the study.
Population: Intent to treat, including all randomized subjects.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control
Number analyzed (Participants) | 432 | 432 | 433
Months | 34.4 [31.0 to 36.9] | 33.2 [30.6 to 37.4] | 34.3 [30.7 to 37.0]
Statistical Analysis 1: Comparison: PROSTVAC-V/F-TRICOM + GM-CSF Placebo vs Placebo Control; Test type: Superiority — One-sided p-value is from a stratified log-rank test for PROSTVAC-V/F-TRICOM + GM-CSF placebo vs. Placebo Control with Treatment Arm included in model. Stratification is by randomization strata; p = 0.4742, Log Rank — The overall type-one error probability for the entire trial was designed as a one-sided P=0.025. There were two main overall comparisons, which necessitated a type-one error probability to 0.0125 for each comparison using a Bonferroni correction; The primary analysis method was a stratified log-rank test, and was performed using the ITT Set analyzing data according to the randomized arm
Statistical Analysis 2: Comparison: PROSTVAC-V/F-TRICOM + GM-CSF vs Placebo Control; Test type: Superiority — One-sided p-value is from a stratified log-rank test for PROSTVAC-V/F-TRICOM + GM-CSF vs. Placebo Control with Treatment Arm included in model. Stratification is by randomization strata; p = 0.5885, Log Rank — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Subjects Alive Without Event at 6 Months
Description: A binary assessment that was performed for the 6-months timepoint for the categories of radiographic progression, pain progression, initiation of chemotherapy or death. Subjects without an event prior to 6-months were evaluated at 6-months. Subjects without event by 6-months and were not evaluated at 6-months were assumed to have had an event and analyzed as such.
  Progression events were defined as: (1) Two new lesions on bone scan, new metastases on CT scans, or an increased size of nodal lesions per RECIST 1.1. Bone or CT scans occurring prior to calendar month 6 were used to determine radiographic progression. (2) Introduction of scheduled opioid narcotics for cancer-related pain control. (3) Initiation of chemotherapy for prostate cancer was assessed as collected on progression forms as well as in cancer treatment and concomitant medications logs. (4) Death.
Time Frame: Randomization through Week 25/End of Treatment visit.
Population: Intent to treat, including all randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control
Number analyzed (Participants) | 432 | 432 | 433
Participants | 127 | 121 | 131
Statistical Analysis 1: Comparison: PROSTVAC-V/F-TRICOM + GM-CSF Placebo vs Placebo Control; Test type: Superiority — Odds Ratio and Wald 95% CI estimates are for odds of alive without event for PROSTVAC-V/F-TRICOM + GM-CSF placebo vs. Placebo Control and are from a logistic regression model with Treatment Arm included in model stratified by randomization strata; Odds Ratio (OR) = 0.9588, 95% CI 2-sided [0.7144 to 1.2867] — The Alive Without Event endpoint was analyzed using stratified logistic regression. The 95% CI on the odds ratio estimate was computed as the measure of the magnitude of effect
Statistical Analysis 2: Comparison: PROSTVAC-V/F-TRICOM + GM-CSF vs Placebo Control; Test type: Superiority — Odds Ratio and Wald 95% CI estimates are for odds of alive without event for PROSTVAC-V/F-TRICOM + GM-CSF vs. Placebo Control and are from a logistic regression model with Treatment Arm included in model stratified by randomization strata; Odds Ratio (OR) = 0.8941, 95% CI 2-sided [0.6647 to 1.2026] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-Emergent AEs were collected from the date of first dose of investigational product through 28 days post-last dose of investigational product, approximately 6 months post-first vaccination for subjects completing the treatment period. All-Cause Mortality was collected for each subject from randomization through death, loss to follow-up, or study closure. Total follow-up lasted approximately 6 years, from the first subject randomized to the completion of the study.
Description: An AE was defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. For the purpose of this clinical trial, AEs included only Treatment-Emergent AEs that were either new or represented detectable exacerbations of pre-existing conditions. Only treated subjects were assessed for adverse events.
Arm/Group | PROSTVAC-V/F-TRICOM + GM-CSF Placebo | PROSTVAC-V/F-TRICOM + GM-CSF | Placebo Control
All-Cause Mortality (participants affected / at risk) | 252/432 | 254/432 | 248/433
Serious Adverse Events (participants affected / at risk) | 56/429 | 56/429 | 53/428
Other Adverse Events (participants affected / at risk) | 351/429 | 367/429 | 346/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROSTVAC-V/F-TRICOM + GM-CSF Placebo (N=429) | PROSTVAC-V/F-TRICOM + GM-CSF (N=429) | Placebo Control (N=428)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2) | 1 (2)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (4) | 7 (8) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 5 (5) | 1 (1) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 4 (4) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular compression (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROSTVAC-V/F-TRICOM + GM-CSF Placebo (N=429) | PROSTVAC-V/F-TRICOM + GM-CSF (N=429) | Placebo Control (N=428)
Constipation (Gastrointestinal disorders) | 39 (44) | 26 (29) | 28 (31)
Diarrhoea (Gastrointestinal disorders) | 38 (41) | 28 (31) | 21 (22)
Nausea (Gastrointestinal disorders) | 51 (65) | 51 (62) | 36 (41)
Asthenia (General disorders) | 32 (46) | 37 (50) | 49 (52)
Chills (General disorders) | 34 (50) | 44 (60) | 35 (42)
Fatigue (General disorders) | 94 (117) | 105 (149) | 91 (116)
Influenza like illness (General disorders) | 44 (68) | 55 (86) | 36 (63)
Injection site erythema (General disorders) | 201 (594) | 256 (765) | 200 (626)
Injection site induration (General disorders) | 46 (98) | 67 (140) | 58 (128)
Injection site oedema (General disorders) | 22 (41) | 23 (47) | 19 (45)
Injection site pain (General disorders) | 109 (252) | 128 (247) | 119 (247)
Injection site pruritus (General disorders) | 77 (145) | 109 (235) | 57 (124)
Injection site swelling (General disorders) | 73 (187) | 101 (247) | 67 (183)
Injection site warmth (General disorders) | 15 (31) | 28 (55) | 21 (38)
Oedema peripheral (General disorders) | 21 (22) | 24 (24) | 12 (12)
Pyrexia (General disorders) | 37 (50) | 91 (142) | 53 (63)
Urinary tract infection (Infections and infestations) | 23 (28) | 17 (22) | 22 (28)
Decreased appetite (Metabolism and nutrition disorders) | 39 (43) | 25 (29) | 31 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (70) | 50 (69) | 55 (71)
Back pain (Musculoskeletal and connective tissue disorders) | 62 (70) | 43 (46) | 48 (55)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 28 (33) | 21 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (46) | 35 (47) | 43 (61)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (34) | 28 (28) | 23 (26)
Dizziness (Nervous system disorders) | 18 (20) | 17 (19) | 22 (25)
Headache (Nervous system disorders) | 32 (67) | 43 (61) | 36 (45)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 20 (24) | 15 (16)
Hot flush (Vascular disorders) | 23 (24) | 20 (21) | 12 (15)
Hypertension (Vascular disorders) | 28 (33) | 23 (26) | 22 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT01322490/SAP_000.pdf
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT01322490/Prot_001.pdf